CLINICAL TRIAL: NCT06826976
Title: Influence of Sensory Electrical Stimulation on Hand Functions in Chronic Stroke Patients
Acronym: SES-Hand
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Hassan Fayed, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/005208
Record Dates: First submitted 2025-02-02; First posted 2025-02-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Hand Functionality
Keywords: stroke; hand function; sensory electrical nerve stimulation; task specific training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: In the context of the study on sensory electrical nerve stimulation (SENS) for chronic stroke patients, a parallel assignment model was utilized. Participants were randomly divided into two groups:
  Study Group (A): Received SENS combined with task-specific training.
  Control Group (B): Received only task-specific training.
  This design facilitated a direct comparison between the two groups to assess the added benefit of incorporating SENS into the rehabilitation program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sensory electrical stimulation (Experimental): received sensory electrical stimulation and task specific training program
  Interventions: Other: sensory electrical stimulation
- Task specific training (Active Comparator): received task specific training program only. Patients were tested pre and post treatment by Grip dynamometer, Pinch dynamometer, Digital goniometer and Action Research Arm Test Scale (ARAT).
  Interventions: Other: task specific training program

INTERVENTIONS:
Other: sensory electrical stimulation — peripheral sensory electrical stimulation on median, ulnar, and radial nerves of affected upper limb, simultaneously with Task Specific Training program which included four subtests of Action Research Arm Test scale.
  Arms: Sensory electrical stimulation
Other: task specific training program — received task specific training program only. Patients were tested pre and post treatment by Grip dynamometer, Pinch dynamometer, Digital goniometer and Action Research Arm Test Scale (ARAT).
  Arms: Task specific training

SUMMARY:
This study investigates the impact of sensory electrical nerve stimulation (SENS) on hand function in chronic stroke patients. Thirty participants were randomly divided into two groups:

Study Group (A): Received SENS combined with task-specific training.

Control Group (B): Received only task-specific training.

Assessments conducted before and after the intervention included measurements of grip strength, pinch strength, wrist range of motion, and performance on the Action Research Arm Test (ARAT).

DETAILED DESCRIPTION:
This study explores the effectiveness of sensory electrical nerve stimulation (SENS) in enhancing hand function among chronic stroke patients. Thirty participants were randomly divided into two groups:

Study Group (A): Received SENS combined with task-specific training.

Control Group (B): Received only task-specific training.

Assessment Methods:

Before and after the intervention, both groups underwent evaluations using:

Grip Dynamometer: To measure grip strength.

Pinch Dynamometer: To assess pinch strength.

Digital Goniometer: To determine wrist flexion and extension range of motion.

Action Research Arm Test (ARAT): To evaluate upper limb functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have experienced their first-ever ischemic stroke in the carotid system domain.
* Age range: 40 to 65 years old.
* Duration of illness: 30 to 180 days since stroke onset.
* Spasticity of the affected hand muscles (wrist flexors, finger flexors, and finger adductors) must be grade 1+ or less according to the Modified Ashworth Scale.
* Hand dysfunction severity ranges from mild to severe, defined by a score of ≤ 4 on the Medical Research Council Scale.

Exclusion Criteria:

* Presence of a deformity in the paralytic upper limb before the stroke.
* History of a lower motor neuron lesion in the impaired upper extremity (e.g., polyneuropathy) before the stroke.
* Skin abrasions or ulcerations on the affected upper limb.
* Unstable health conditions, including cardiac dysfunction, end-stage renal failure, unstable diabetes, or uncontrolled hypertension (>190/110).
* Presence of a pacemaker or other implanted electrically sensitive devices.
* Significant orthopedic conditions or chronic pain syndromes.
* Chronic use of medications that may influence motor or sensory excitability (e.g., anti-epileptic or antipsychotic drugs).
* Pregnancy.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | From enrollment to the end of treatment at end of 4th week
  The patient seated with his/her shoulder adducted and naturally rotated, elbow flexed at 90 degrees, forearm in neutral position, and wrist between 0- and 30-degrees dorsiflexion and between 0- and 15-degrees ulnar deviation. The Jamar hand dynamometer was set to the second handle position from the inside. Lightly hold around the readout dial to prevent inadvertent dropping. After the patient was positioned properly, the following statement was used "Squeeze as hard as you can…. harder …. harder…. relax" (16). The scores of three successive trials were recorded for each tested hand. The average score of three trials was compared to the normative data on the other side, which is in pounds.
wrist range of motion | From enrollment to the end of treatment at end of 4th week
  Goniometer was used to assess wrist flexion-extension.
pinch strength | From enrollment to the end of treatment at end of 4th week
  Three types of pinches were typically evaluated because they are involved in accomplishing occupational tasks and activities efficiently. In Tip Pinch: The patient pinched the ends of the pinch meter between the tips of the thumb and index finger. The test was administered by first giving the patient instructions and a demonstration, "Ready? Pinch as hard as you can." The patient was urged on as he or she attempted to pinch. The average of three trials was recorded. In Lateral Pinch (Key Pinch): The patient pinched the meter between the pad of the thumb and the lateral surface of the index finger. In Palmar Pinch (Three-Jaw Chuck): The patient pinched the meter between the pad of the thumb and the pads of the index and middle fingers
hand functions | From enrollment to the end of treatment at end of 4th week
  Patients who achieve a maximum score on the first (most difficult) item are credited with having scored 3 on all subsequent items on that scale. If the patient scores less than 3 on the first item, then the second item is assessed. This is the easiest item, and if patients score 0 then they are unlikely to achieve a score above 0 for the remainder of the items and are credited with a zero for the other items. The maximum score on ARTS is 57 points (possible range 0 to 57).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided